CLINICAL TRIAL: NCT07272395
Title: Monitoring Right Ventricular Function in Patients Undergoing Implantable Cardiac Electronic Device (CIED) Therapy: A Multimodal Imaging and Biomarker-Based Approach
Brief Title: Right Ventricular Function Changes After CIED Implantation: The RIGHT-CIED Study
Acronym: RIGHT-CIED
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sahra Asena Balcioglu, Resident Physician, Cardiology Department, Istanbul University - Cerrahpasa
Other Study IDs: 2025/619IUCIC
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-08

CONDITIONS: Right Ventricular Dysfunction
Keywords: right ventricular dysfunction; right ventricular function; Cardiac Implantable Electronic Device; Implantable Cardioverter-Defibrillator; pacemaker; Cardiac Resynchronisation Therapy; Cardiac Magnetic Resonance Imaging; Echocardiography; VExUS; Venous Congestion; Fibroblast Growth Factor 23; Brain Natriuretic Peptide
MeSH Terms: conditions — Ventricular Dysfunction, Right; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — EDTA plasma samples derived from venous whole blood; stored for biomarker analysis (FGF-23 and BNP). No DNA extraction will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIED Implantation Cohort: Participants with an indication for the implantation of an implantable cardiac electronic device (pacemaker, ICD, or CRT) as part of routine clinical care. All participants will undergo detailed assessment of right ventricular structure and function immediately before device implantation and again at 6 months after implantation. Assessments include transthoracic echocardiography, VEXUS ultrasound scoring, non-contrast cardiac MRI, and blood sampling for biomarker analysis (FGF-23 and BNP). No experimental intervention is administered; all implanted devices are clinically indicated.
  Interventions: Other: Multimodal Right Ventricular Evaluation

INTERVENTIONS:
Other: Multimodal Right Ventricular Evaluation — Non-invasive assessments including transthoracic echocardiography, VEXUS ultrasound scoring, non-contrast cardiac MRI using 1.5T scanner, and venous blood sampling for EDTA plasma biomarker analysis (FGF-23 and BNP). These procedures are for research measurements only and do not alter or replace routine clinical care. No therapeutic intervention or assignment is performed.

SUMMARY:
This study aims to understand how the right side of the heart changes in people who receive an implantable cardiac electronic device (CIED), such as a pacemaker, ICD, or CRT device. The right ventricle (RV) can sometimes be affected after these devices are placed, but the reasons and timing are not well understood.

To investigate this, we will examine participants at two time-points: before their device is implanted and again six months later. At each visit, we will assess heart function using echocardiography, a non-contrast cardiac MRI scan, and an ultrasound score of venous congestion called the VEXUS score. We will also take a small blood sample to measure a biomarker called FGF-23, which may reflect changes in heart function.

The study does not involve any experimental treatment, and all implanted devices are part of routine medical care. The imaging tests and blood samples are for research purposes only. By comparing the measurements before and after device implantation, we hope to better understand how CIEDs influence right-sided heart function and whether imaging findings are related to changes in blood biomarkers.

DETAILED DESCRIPTION:
Right ventricular (RV) dysfunction and tricuspid valve changes are increasingly recognised in patients who receive implantable cardiac electronic devices (CIEDs). Potential mechanisms include lead-leaflet interaction, pacing-related alterations in RV mechanics and changes in venous haemodynamics. However, prospective data integrating advanced imaging, ultrasound-based congestion assessment and circulating biomarkers remain limited.

This prospective observational cohort study will evaluate RV structure and function at two predefined time-points: immediately before CIED implantation and at six months after implantation. Assessments will include (1) transthoracic echocardiography with quantitative RV parameters, (2) a standardised VEXUS ultrasound score for systemic venous congestion, (3) non-contrast cardiac magnetic resonance (CMR) imaging for RV volumetry and tissue characterisation and (4) plasma measurement of FGF-23 as a biomarker potentially associated with RV remodelling.

All implanted devices are clinically indicated and form part of routine care; no experimental device or therapeutic intervention is used. Imaging and blood sampling performed for the study are non-interventional and carry minimal risk. The purpose of the study is to quantify changes in RV size and function over six months and to explore whether alterations in imaging findings correspond to changes in venous congestion or biomarker levels. The results may help identify patients at risk of adverse RV remodelling following CIED implantation.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older.
* Scheduled to undergo implantation of a clinically indicated pacemaker, ICD, or CRT device.
* Able to undergo transthoracic echocardiography, VEXUS ultrasound assessment, and non-contrast cardiac MRI.
* Able to provide written informed consent.

Exclusion Criteria

* Contraindication to cardiac MRI (e.g., severe claustrophobia or MRI-unsafe implanted material).
* Inability to undergo echocardiography or ultrasound assessment.
* Known pulmonary arterial hypertension (Group 1 PH).
* Significant congenital heart disease.
* Patients with mechanical or bioprosthetic heart valve replacement
* Severe left-sided valvular disease (severe AS or severe MR).
* Chronic kidney disease stage 4 or 5 (eGFR < 30 mL/min/1.73m²).
* End-stage renal disease requiring dialysis.
* Primary hyperparathyroidism.
* Hypophosphataemia or hyperphosphataemia requiring treatment.
* Active or uncontrolled bone metabolism disorders (e.g., osteomalacia, Paget's disease).
* Recent fracture or major orthopaedic surgery within the past 3 months.
* Active systemic inflammatory or autoimmune disease.
* Active malignancy or malignancy requiring ongoing treatment.
* Active infection at the time of enrolment.
* Pregnancy or breastfeeding.
* Haemodynamic instability at the time of enrolment.
* Expected survival less than 6 months due to non-cardiac conditions.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the cardiology clinics and electrophysiology unit of Istanbul University-Cerrahpaşa Cardiology Institute. The study population consists of adult patients scheduled for implantation of a clinically indicated pacemaker, ICD, or CRT device. All participants represent a routine tertiary-care population referred for device therapy due to bradyarrhythmia, heart failure, or ventricular arrhythmia indications.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Change in Right Ventricular Ejection Fraction (RVEF) by Cardiac MRI | Baseline (pre-implantation) to 6 months post-implantation
  RVEF will be quantified using non-contrast 1.5T cardiac MRI cine imaging. The primary endpoint is the absolute change in RVEF between pre-implantation and 6-month follow-up.
Change in Tricuspid Regurgitation Severity | Baseline to 6 months
  Tricuspid regurgitation will be graded (none, mild, moderate, severe) using echocardiography and confirmed by CMR-derived regurgitant volume.

SECONDARY OUTCOMES:
Change in Right Ventricular End-Diastolic Volume (RVEDV) by Cardiac MRI | Baseline to 6 months
  RVEDV will be measured from short-axis cine stacks. The endpoint is the change in volume between baseline and 6 months.
Change in VEXUS Score | Baseline to 6 months
  VEXUS venous congestion score (IVC, hepatic vein Doppler, portal vein pulsatility, renal vein Doppler) will be calculated at each visit.
Change in Right Ventricular Longitudinal Strain (RV-FWLS) | Baseline to 6 months
  Measured via speckle-tracking echocardiography.
Change in Plasma FGF-23 Concentration | Baseline to 6 months
  EDTA plasma FGF-23 will be measured via ELISA. The endpoint is the change in concentration from baseline to 6 months.
Change in BNP Concentration | Baseline to 6 months
  Plasma BNP levels will be measured as a secondary biochemical marker.
Lead-related Tricuspid Valve Interaction | 6 months
  Based on CMR evaluation of lead-leaflet relationship (septal, posteroseptal, anterior leaflet proximity or impingement).

CONTACTS AND LOCATIONS:
Overall Officials: SAHRA ASENA BALCIOGLU, Principal Investigator — ISTANBUL UNIVERSITY-CERRAHPASA INSTITUTE OF CARDIOLOGY
Locations (1):
- Istanbul University-Cerrahpasa Institute of Cardiology, Istanbul, FATIH, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to right ventricular measurements, echocardiographic parameters, VEXUS scores, cardiac MRI-derived volumetric results, and biomarker values (FGF-23 and BNP) may be shared. No direct identifiers, imaging files, or raw MRI data will be provided. Only anonymised numerical data used for statistical analysis will be available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be available from 12 months to 5 years after publication.
Access Criteria: De-identified individual participant data (IPD) will be accessible to qualified researchers affiliated with recognised academic or clinical institutions. Access will be granted for the purpose of scientific analysis only, upon submission of a reasonable research proposal and approval by the study investigators. Data will be shared in an anonymised electronic format via secure data transfer. No identifiable information, imaging files, or raw MRI datasets will be provided.

REFERENCES:
- [Result] Zoghbi WA, Addetia K, Bhave PD, et al. Tricuspid Regurgitation in Patients With Cardiac Implantable Electronic Devices: JACC Scientific Expert Panel. J Am Coll Cardiol. 2023;82(13):1284-1302. PMID: 37708963
- [Result] Benes J, Kroupova K, Kotrc M, Petrak J, Jarolim P, Novosadova V, Kautzner J, Melenovsky V. FGF-23 is a biomarker of RV dysfunction and congestion in patients with HFrEF. Sci Rep. 2023 Sep 25;13(1):16004. doi: 10.1038/s41598-023-42558-4. PMID 37749114